CLINICAL TRIAL: NCT01682551
Title: Evaluation of the Prevention and Treatment Effects of Chinese Medicine on High Altitude Illness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NRICM-10101
Record Dates: First submitted 2012-09-05; First posted 2012-09-11 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Acute Mountain Sickness (AMS)
Keywords: High altitude illness; Chinese medicine body constitution; Chinese Medicine; High altitude medicine; Mountain trekking
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chinese Medicine (Experimental): The participators in this arm will take 2g (powder in capsule) of "Wu Zhu Yu Tang" or placebo orally three times in the first day and one time in the second day.
  Interventions: Drug: Chinese Medicine
- Acetazolamide (Placebo Comparator): If the participators have the history of AMS, he/she will be randomized to take "Wu Zhu Yu Tang" plus "placebo of Acetalozamide" or "Acetalozamide" plus "placebo of Wu Zhu Yu Tang".
  Interventions: Drug: Chinese Medicine; Drug: Acetalozamide

INTERVENTIONS:
Drug: Chinese Medicine — The participators in this arm will take 2g (powder in capsule) of "Wu Zhu Yu Tang" or placebo orally three times in the first day and one time in the second day.
  Other Names: "Wu Zhu Yu Tang"
Drug: Acetalozamide — If the participators have the history of AMS, he/she will be randomized to take "Wu Zhu Yu Tang" plus "placebo of Acetalozamide" or "Acetalozamide" plus "placebo of Wu Zhu Yu Tang".
  Arms: Acetazolamide

SUMMARY:
This trial is aimed to evaluate the effects of "Wu Zhu Yu Tang" on the prevention of Acute Mountain Sickness(AMS).

DETAILED DESCRIPTION:
This study is a randomized, double blind, placebo-controlled clinical trial. It aims to demonstrate that (1) Chinese medicine prescription "Wu Zhu Yu Tang" can prevent Acute Mountain Sickness(AMS) (2) "Wu Zhu Yu Tang" can prevent AMS especially for Yang-Xu body constitution.

We will randomize 240 unacclimatized healthy adults. They will be randomized after stratification of the Yang-Xu score and the AMS history to receive Chinese medicine during one ascent and placebo during the other ascent. We will take them in Hehuan mountain for two days hike (24 hours) and an overnight over 3,000m. One month before the study, the subjects will fill the "Body Constitution Questionnaire BCQ" in order to evaluate their body constitution. Before, during and after the two days hike we will measure their blood pressure, heart rate and arterial oxygen saturation. The incidence of AMS will be measured by the Lake Louise Self Report (Lake Louise Score ≥4 with headache), we will also report the Lake Louise Clinical Assessment score and Lake Louise Functional Score.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Chronic disease: cardiovascular disease, psychological disease, anemia, migraine.
* long-term use of the following materials: Chinese herbs, steroid, antibiotics.
* altitude acclimation: have been to mountain over 2000m in the past 1 month.
* Pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of AMS will be measured by the Lake Louise Self Report (Lake Louise Score ≥4 with headache) | The Lake Louise Score will be measured in the noon of the second day after hiking to determine the onset of AMS.
  The investigators will take the participators in Hehuan mountain for two days hike (24 hours) and an overnight over 3,000m. The Lake Louise score will measure before and after hiking.

SECONDARY OUTCOMES:
Blood pressure | Blood pressure will be measured before and after the hiking.
  The investigators will take the participators in Hehuan mountain for two days hike (24 hours) and an overnight over 3,000m. The change of blood pressure will be measured before and after hiking.
Heart rate | Heart rate will be measured before and after the hiking.
  The investigators will take the participators in Hehuan mountain for two days hike (24 hours) and an overnight over 3,000m. The change of heart rate will be measured before and after hiking.
Arterial oxygen saturation | Arterial oxygen saturation will be measured before and after the hiking.
  Description:
  The investigators will take the participators in Hehuan mountain for two days hike (24 hours) and an overnight over 3,000m. The change of arterial oxygen saturation will be measured before and after hiking.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Chinese Medicine, China Medical University, Taichung, Taiwan, Taiwan